CLINICAL TRIAL: NCT06867419
Title: Metabolic Features Effect on FibroScan-AST (FAST) Score in Egyptian Patients With Metabolic-Associated Steatotic Liver Disease (MASLD)
Brief Title: Metabolic Features Effects on FAST Score in MASLD Patients
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Lecturer of Tropical medicine, Tanta University
Other Study IDs: 36264PR889/10/24
Record Dates: First submitted 2025-02-13; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: Metabolic dysfunction-Associated Steatotic Liver Disease (MASLD); FAST Score; Metabolic Features

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MASLD patients: 385 MASLD patients who had steatosis detected by (VCTE-CAP) elastography
  Interventions: Radiation: Transient Elastography

INTERVENTIONS:
Radiation: Transient Elastography — participants will be subjected to anthropometric measurements, laboratory investigations (complete blood count, liver and kidney functions, lipid profile, virology tests, fasting insulin, fasting sugar, 2 hour postprandial sugar, HbA1c, and HOMA-IR), radiological examination (abdominal ultrasound, Fibroscan). the NAFLD fibrosis score, APRI, FIB-4 score, and FAST score will be calculated.

SUMMARY:
The goal of this observational cross-sectional study is to evaluate the effect of metabolic features on Fibroscan-AST (FAST) score stratification in metabolic dysfunction-associated steatotic liver disease (MASLD) patients in Egypt.

Researchers will identify the metabolic risk factors in patients with MASLD. evaluate the effect of metabolic features on stratifying MASLD patients by predicting higher FAST score.

Participants will be subjected to history taking, clinical examination, laboratory investigations, abdominal ultrasonography, and transient elastography (Fibroscan) to measure liver stiffness (LSM) and controlled attenuation parameter (CAP). The Non-alcoholic fatty liver disease (NAFLD) fibrosis score and FAST score will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* All patients with MASLD who had steatosis detected by (VCTE-CAP) elastography

Exclusion Criteria:

* Patients with a history of significant alcohol consumption more than 30 g/day in men and > 20 g/day in women.
* Patients with positive hepatitis B or C virus markers.
* Patients with autoimmune hepatitis.
* Patients with any other metabolic liver disease.
* Patients with hepatic focal lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects from the outpatient clinic of the Tropical Medicine and Infectious Diseases Department at Tanta University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
impact of metabolic features on FAST score | through study completion, an average of 6 months
  Calculating the FAST score by combining AST (IU/L) with LSM (kPa) and CAP (dB/m2) measured by Fibroscan for all MASLD patients. Evaluation of which metabolic features (DM, HTN, obesity, dyslipidemia) would be associated with a higher FAST score indicating having steatohepatitis with significant inflammatory activity and fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Rania M Elkafoury, MD, Study Director — Tropical medicine and infectious diseases Department, Faculty of Medicine, Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Gharbyea, Egypt